CLINICAL TRIAL: NCT06358170
Title: Effects of Circuit Training Combine With Square-Stepping Exercise, Strength Training and Balance Training on Senior Fitness and Fall Risk in Elderly in the Community
Acronym: SSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hsin-ching, Tsai (Other)
Responsible Party: Sponsor-Investigator, Hsin-ching, Tsai, Student, National Yang Ming Chiao Tung University
Organization: National Yang Ming Chiao Tung University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NYCU112169AF
Record Dates: First submitted 2024-03-24; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Circuit-Based Exercise; Exercise Test; Community Health Nursing; Aged; Physical Fitness
Keywords: community; elderly people; falls; fall prevention; Square-Stepping Exercise; circuit training; exercise training; physical fitness; cognitive function; fear of falling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSE (Experimental): A Circuit Training Combine with Square-Stepping Exercise, Strength training and balance training. The intervention time and frequency of this study were 12 weeks, 2 times a week, 24 times in total, 1.5 hours each time (30 minutes of main exercise).
  Interventions: Behavioral: Circuit Training Combine with Square-Stepping Exercise
- Control (No Intervention): No intervention (daily routine)

INTERVENTIONS:
Behavioral: Circuit Training Combine with Square-Stepping Exercise — Circuit Training Combine with Square-Stepping Exercise
  Arms: SSE

SUMMARY:
According to the cause of death statistics compiled by the Ministry of Health and Welfare in 2022, among the causes of death among the elderly, falls ranked second among the causes of death from accidental injuries over the age of 65. Exercise has been proven to prevent falls in many studies, especially Square-Stepping Exercise can not only train strength and balance, but also improve cognitive function and reduce the fear of falling in the elderly. Therefore, this study will use Square-Stepping Exercise as the core and circuit training as the structure to design a set of exercise training that combines muscle strength and balance and is easy to implement in the community. The purpose of the study is to determine whether exercise training that combines circuit training with block stepping, muscle strength, and balance exercises can reduce the risk of falls among elderly people in the community (primary results: muscle strength, flexibility, cardiorespiratory endurance, balance; secondary results: cognitive function, Fear of falling, fall rate). This study will collect participant in the community, and subjects will be randomly assigned to the experimental group and the control group on a community basis. The experimental group will receive 12 weeks of exercise training, while the control group will follow their usual lifestyle, with 48 people in each group. The experimental design is exercise intervention for 12 weeks, twice a week, 90 minutes each time (30 minutes of main exercise). The exercise is designed into two stages according to the difficulty of Square-Stepping Exercise. The training of muscle strength and dynamic/static balance will also gradually increase in difficulty over the weeks. The research look forward to seeing the effects of multi-component exercise on physical fitness, cognitive function, fear of falling and fall rate.

DETAILED DESCRIPTION:
With the improvement of medical and sanitation, the average life expectancy of human beings around the world has gradually increased, which has led to the trend of an aging society. Therefore, the health issues of the elderly have received more attention. Aging should cause impairment of human body functions, including significant decline in sensory systems (vision, hearing, vestibular, proprioception, etc.), muscle strength, muscle endurance, balance, and gait functions, which may increase accidental falls or injuries. risks. According to the cause of death statistics compiled by the Ministry of Health and Welfare in 2022, among the causes of death among the elderly, falls ranked second among the causes of death from accidental injuries over the age of 65. According to the literature, it was found that most of the causes of falls among the elderly are related to internal factors (including decreased muscle strength, balance, and cognitive function), and exercise has been proven to prevent falls in many studies, especially Square-Stepping Exercise can not only train strength and balance, but also improve cognitive function and reduce the fear of falling in the elderly. It is an intervention method that is easy to implement in the community. Compared with traditional resistance training, circuit training is shorter duration and lower intensity, which may increase compliance with training assistance. Also, can make up for shortcomings of Square-Stepping Exercise. Training takes turns, resulting in long waiting times for a class. In experiments on exercise intervention, it was found that multicomponent exercise combined with a variety of exercises is more effective in preventing falls than a single type of exercise. Therefore, this study will use Square-Stepping Exercise as the core and circuit training as the structure to design a set of exercise training that combines muscle strength and balance and is easy to implement in the community. The purpose of the study is to determine whether exercise training that combines circuit training with block stepping, muscle strength, and balance exercises can reduce the risk of falls among elderly people in the community (primary results: muscle strength, flexibility, cardiorespiratory endurance, balance; secondary results: cognitive function, Fear of falling, fall rate). This study will collect participant in the community, and subjects will be randomly assigned to the experimental group and the control group on a community basis. The experimental group will receive 12 weeks of exercise training, while the control group will follow their usual lifestyle, with 48 people in each group. The experimental design is exercise intervention for 12 weeks, twice a week, 90 minutes each time (30 minutes of main exercise). The exercise is designed into two stages according to the difficulty of Square-Stepping Exercise. The training of muscle strength and dynamic/static balance will also gradually increase in difficulty over the weeks. The research data were analyzed using IBM SPSS, and we look forward to seeing the effects of multi-component exercise on physical fitness, cognitive function, fear of falling and fall rate.

Keywords: community, elderly people, falls, fall prevention, Square-Stepping Exercise, circuit training, exercise training, physical fitness, cognitive function, fear of falling

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 years or older.
2. Determine no exercise risk via ACSM's PAR-Q+ (The Physical Activity Readiness Questionnaire for everyone).
3. SPPB (Short Physical Performance Battery) score of 10 or above indicates normal mobility.
4. Will not participate in other physical exercise programs after starting this program.

Exclusion Criteria:

1. Those who are unable to complete the assessment process (due to hearing, vision, etc.) or participate due to limited mobility problems.
2. Those whose cognitive function cannot cooperate with the assessment process.
3. Those whose attendance rate is less than 80%.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Senior Fitness - upper body muscle strength (Arm Curl Test) | 30 seconds
  As the arm is lowered through the full range of motion, gradually return to the starting position. The arm must be fully bent and then fully straightened at the elbow. Repeat this action as many times as possible within 30 seconds.
Senior Fitness - lower body muscle strength (Chair Stand Test ) | 30 seconds
  From the sitting position, the subject stands completely up, then completely back down, and this is repeated for 30 seconds. Count the total number of complete chair stands (up and down equals one stand).
Senior Fitness - upper body flexibility (Back Scratch Test) | 5 seconds
  Place one hand behind the head and back over the shoulder, and reach as far as possible down the middle of your back, your palm touching your body and the fingers directed downwards. Place the other arm behind your back, palm facing outward and fingers upward and reach up as far as possible attempting to touch or overlap the middle fingers of both hands. An assistant is required to direct the subject so that the fingers are aligned, and to measure the distance between the tips of the middle fingers. If the fingertips touch then the score is zero. If they do not touch, measure the distance between the finger tips (a negative score), if they overlap, measure by how much (a positive score).
Senior Fitness - lower body flexibility (Chair Sit and Reach Test) | 5 seconds
  The subject should sit on the edge a chair (placed against a wall for safety). One foot must remain flat on the floor. The other leg is extended forward with the knee straight, heel on the floor, and ankle bent at 90°. Place one hand on top of the other with tips of the middle fingers even. Keep the knee straight, and hold the reach for 2 seconds. The distance is measured between the tip of the fingertips and the toes. If the fingertips touch the toes then the score is zero. If they do not touch their toes, measure the distance between the fingers and the toes (a negative score), if they overlap, measure by how much (a positive score). Perform two trials.
Senior Fitness - cardio respiratory endurance ( 2 Minute Step in Place Test) | 2 minutes
  The subject stands up straight next to the wall while a mark is placed on the wall at the level corresponding to midway between the patella (knee cap) and illiac crest (top of the hip bone). The subject then marches in place for two minutes, lifting the knees to the height of the mark on the wall. Stop after two minutes of stepping.
Senior Fitness - dynamic balance (8-Foot Up and Go Test) | 10 seconds
  Place the chair next to a wall (for safety) and the marker 8 feet in front of the chair. Clear the path between the chair and the marker. The subject starts fully seated, hands resting on the knees and feet flat on the ground. On the command, "Go," timing is started and the subject stands and walks (no running) as quickly as possible (and safely) to and around the cone, returning to the chair to sit down. Timing stops as they sit down. Perform two trials.
Senior Fitness - static balance (Single-Leg Balance with Eyes Open) | 30 seconds
  Performed with eyes open and hands on the hips. Stands on one leg unassisted; time begins when opposite foot leaves the ground; time stops immediately when opposite foot touches the ground and/or when hands leave the hips. 30 seconds is the best time, if it exceeds 30 seconds, it will be scored as 30 seconds.

SECONDARY OUTCOMES:
cognitive function | 7 minutes
  The Saint Louis University Mental Status Examination (SLUMS)
Fear of falling | 2 minutes
  The Falls Efficacy Scale-International (FES-I)
fall rate | 30 seconds
  Number of falls and trips in the past 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided